CLINICAL TRIAL: NCT01489163
Title: Translational Diabetes Prevention in GDM
Brief Title: Lifestyle Intervention Program for Women With Gestational Diabetes or Gestational Impaired Glucose Tolerance
Acronym: APPLES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CN-03AFerr-02-H
Record Dates: First submitted 2011-12-07; First posted 2011-12-09 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Gestational Diabetes
Keywords: Gestational Diabetes; Weight Loss; Physical Activity; Pregnancy; Postpartum; Intervention
MeSH Terms: conditions — Diabetes, Gestational; Weight Loss; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle Counseling (Experimental)
  Interventions: Behavioral: Lifestyle Counseling
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Lifestyle Counseling — The Phase I intervention will be delivered through 1 individual in-person session and 3 individual telephone counseling contacts. The Phase II intervention begins at 6-week postpartum and will be delivered through 3 individual in-person sessions and 13 telephone counseling contacts over a period of 6 months. The maintenance phase (Phase III) will begin at 8 months postpartum.
  Arms: Lifestyle Counseling

SUMMARY:
The purpose of this research study is to implement and evaluate a lifestyle program designed to help women who have high glucose levels during pregnancy make healthful diet and physical activity changes to lose weight. Eligible women will be randomly assigned to life-style intervention or usual medical care.

ELIGIBILITY:
Inclusion Criteria:

* Women receiving prenatal care at Kaiser Permanente Santa Clara, Santa Teresa, Hayward, and Oakland
* Pregnancy complicated by high glucose levels starting November 2011

Exclusion Criteria:

* Recognized DM prior to pregnancy
* Uncontrolled hypertension during pregnancy
* Severe active thyroid disease during pregnancy
* Severe diseases of the cardio-pulmonary system
* Diagnosis of a severe psychiatric disorder
* Diagnosis of cancer
* Conditions that lead to diet changes
* Addiction to alcohol or illegal drugs
* Current corticosteroid medicine use

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 352 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
postpartum body weight | through 24 months postpartum

SECONDARY OUTCOMES:
the proportion of women who reach body weight goals | through 24 months postpartum
percent of calories from fat | through 24 months postpartum
time spent in physical activity (PA) by intensity | through 24 months postpartum
postpartum glycemia | through 24 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Assiamira Ferrara, MD, PhD, Principal Investigator — Kaiser Permanente Division of Research
Locations (1):
- Division of Research Northern California, Oakland, California, United States